CLINICAL TRIAL: NCT03612778
Title: Nutritional Intervention for Management of Cardiovascular Risk Factors in Kidney Transplant Patients
Brief Title: Modification of Diet in Renal Transplantation (MDRT)
Acronym: MDRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Jernej Pajek, Professor Jernej Pajek, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MDRT
Record Dates: First submitted 2018-06-28; First posted 2018-08-02 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Kidney Transplant; Complications
Keywords: nutrition; dyslipidemia; insulin resistance; inflammation
MeSH Terms: conditions — Dyslipidemias; Insulin Resistance; Inflammation | interventions — Diet, Plant-Based; Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two parallel groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant-based diet (Experimental): Participants will receive a meal plan based on unrefined plant-based foods with the following macronutrient composition: approximately 15% of calories from vegetable protein, <15% from fat, and 70-75% from carbohydrates. Additionally, to ensure adequate intake of n-3 polyunsaturated fatty acids, they will receive a supplement in the form of one 840 mg n-3 acids eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) daily. Nutritional intervention includes dietary counselling and weekly peer-group meetings together with a next of kin.
  Interventions: Behavioral: Plant-based diet
- Mediterranean diet (Active Comparator): Participants will receive a meal plan, based on the recommendations by the Task Force for the Management of Dyslipidaemias of the European Society of Cardiology and European Atherosclerosis Society, based on Mediterranean diet pattern with the following macronutrient composition: approximately 15% of calories from animal and vegetable protein, up to 30% of calories from fat, 50-65% from carbohydrates. Nutritional intervention includes dietary counselling and weekly peer-group meetings together with a next of kin.
  Interventions: Behavioral: Mediterranean diet

INTERVENTIONS:
Behavioral: Plant-based diet — Prescription of a meal plan based on unrefined plant-based foods supported by peer group meetings and dietary counselling. Change from the standard western-type nutritional pattern to a low-fat, unrefined, plant-based nutritional pattern.
  Arms: Plant-based diet
Behavioral: Mediterranean diet — Prescription of a meal plan based on Mediterranean diet pattern supported by peer group meetings and dietary counselling. Change from the standard western-type nutritional pattern to a Mediterranean nutritional pattern.
  Arms: Mediterranean diet

SUMMARY:
Abnormalities in lipid metabolism are present in 50-80% of patients with a kidney transplant and together with concurrent comorbidities and other associated cardiovascular risk factors put kidney transplant recipients at a high-risk for cardiovascular disease. First line lipid-lowering therapy in this population is pharmacological with 3-hydroxy-3-methyl-glutaryl-coenzyme A (HMG-CoA) reductase inhibitors (statins), however there is a paucity of data on the efficacy of therapeutic lifestyle modification for cardiovascular risk management in kidney transplant recipients. The aim of the present study is to assess efficacy, safety and feasibility of a nutritional intervention for lowering cardiovascular risk factors in kidney transplant recipients. Investigators will conduct a randomized controlled trial on the effects of a low-fat, unrefined, plant-based diet compared to the currently recommended diet according to nutrition guidelines and based on the Mediterranean diet pattern to lower the primary end-point LDL-cholesterol and other secondary end-points validated as risk factors for cardiovascular events. Length of the intervention will be 6 weeks, with a late follow-up after additional 3 months. Stabile kidney transplant recipients with LDL-cholesterol >2.6 mmol/l and/or receiving lipid lowering treatment will be randomized in a 1:1 ratio to either interventional low-fat, unrefined, plant-based diet or to a control diet based on the Mediterranean dietary pattern. Both diets will be prescribed in the form of a weekly menu, both will be allowed to be eaten ad libitum (without prespecified calorie restriction) and in both groups study participants will be supported by tutor classes and counseling to maximise their adherence to prescribed dietary pattern.

DETAILED DESCRIPTION:
BACKGROUND. Abnormalities in lipid metabolism are present in 50-80% of patients with a kidney transplant, as a consequence of both the primary cause of end-stage renal disease, its complications and immunosuppressive therapy. Concurrent comorbidities and cardiovascular risk factors put kidney transplant recipients at high-risk for cardiovascular disease, therefore the target LDL-cholesterol was set to below 2.6 mmol/l (< 100 mg/dl) by the guidelines. First line lipid-lowering therapy in this population is pharmacological, namely with HMG-CoA reductase inhibitors (statins), which have potential interactions with immunosuppressive drugs and increased risk of adverse effects. There is a paucity of data on the efficacy of therapeutic lifestyle modification for cardiovascular risk management in the kidney transplant recipient. Studies in the general population showed a significant effect of mostly plant-based nutrition on lowering lipid levels, achieving approximately 10-15% reduction in both total and LDL-cholesterol, while the effect on cardiovascular protection of such nutritional intervention remains hypothetical. The aim of the present study is to confirm efficacy, safety and feasibility of nutritional intervention for lowering cardiovascular risk factors in kidney transplant recipients. METHODS. Investigators will conduct a randomized controlled trial on the effects of a low-fat, unrefined, plant-based diet compared to the currently recommended diet based on the Mediterranean dietary pattern and complying with current nutrition guidelines for general population to lower LDL-cholesterol. Duration of dietary intervention will be 6 weeks with further extension of intervention and assessment of end-points after additional 3 months. Final follow-up is scheduled after 12 months regardless of continuation of the intervention as decided by subjects themselves. Subjects in the experimental group will receive a meal plan based on low-fat, unrefined, plant based foods with the goal macronutrient intake of approximately 15% protein, <15 % fats and 70-75% of carbohydrates, and will additionally receive polyunsaturated fatty acid (PUFA n-3) supplement (daily dose 840 mg) to ensure daily recommended intake. Subjects in the control group will receive a meal plan in accordance with recommendations by the Task Force for the Management of Dyslipidaemias of the European Society of Cardiology and European Atherosclerosis Society incorporating foods according to the Mediterranean dietary pattern including the usage of (but not limited to) olive oil, fatty-fish and low-fat dairy products. To promote adherence to the meal plan, subjects will receive dietary counselling and will be invited to attend weekly peer-group meetings together with a next of kin. Both diets will be allowed to be eaten at libitum and no calorie counts will be made. A random 24-hour recall, announced prospective 3-day food diary analysis and analysis of a 24-hour urine collection to determine adherence to the prescribed meal plan will be performed. To ensure safety, periodically monitoring of basic serum electrolyte concentrations, body weight and composition, and adjustment of antihypertensive and antihyperglycemic medications will be allowed. No change of lipid lowering agents will be allowed for the first 6-week study period. Feasibility of the intervention will be assessed by adherence monitoring as described above and with the Kidney Disease Quality of Life Short Form questionnaire. Analysis of covariance with baseline parameter value used as a covariate will be used for primary statistical analysis. Based on expected effect of nutritional intervention on lowering LDL-cholesterol by 0.6 mmol/l (23 mg/dl) in the study population by the end of intervention period, standard deviation of LDL-cholesterol of 0.6 mmol/l (23 mg/dl) in the study population with the expected drop-out rate of 15 %, the required sample size of 43 participants in each group to achieve a statistical significance p < 0.05 and statistical power of 80% is defined.

ELIGIBILITY:
Inclusion Criteria:

* recipient of kidney transplant > 12 weeks after transplantation and evaluated as clinically stable
* age 18 years or more at inclusion
* estimated glomerular filtration rate (GFR) > 15 ml/min/1.73
* diagnosed dyslipidemia (LDL-cholesterol > 2.6 mmol/l (> 100 mg/dl) at inclusion or receiving lipid-lowering therapy)
* ability to participate in a lifestyle modification study.

Exclusion Criteria:

* acute illness, infection or surgical intervention requiring hospitalization in 6 weeks before inclusion, except procedures relating to arteriovenous fistula
* treatment of acute rejection or citomegalovirus infection in 6 weeks before inclusion
* chronic illness, associated with or increasing the risk of cachexia (including congestive heart failure New York Heart Association III or IV, AIDS, advanced chronic obstructive pulmonary disease, metastatic neoplastic disease or locally active neoplastic disease, chemotherapy treatment in 6 weeks before inclusion)
* clinically evident malnutrition (BMI < 18,5, reduction of body weight > 5% in 3 months before inclusion, reduction of dietary intake > 25 % from normal in 2 weeks before inclusion, serum albumin < 30 g/l (< 3 g/dl))
* nephrotic syndrome
* pregnancy
* treatment with vitamin K antagonists
* change in lipid-lowering therapy in 3 weeks before inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2018-11-15 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Serum low density lipoprotein (LDL)-cholesterol | 6 weeks and 3 months
  Serum LDL-cholesterol concentration

SECONDARY OUTCOMES:
Apolipoprotein B | 6 weeks and 3 months
  Apolipoprotein B serum concentration
Reduction in insulin resistance | 6 weeks and 3 months
  Change in insulin resistance, measured by Homeostatic Model Assessment (HOMA-IR)
Serum cholesterol | 6 weeks and 3 months
  Serum total cholesterol concentration
Oxidized Low Density Lipoprotein (LDL)-cholesterol | 6 weeks and 3 months
  Serum concentration of oxidized LDL-cholesterol
Inflammatory marker high sensitive C-Reactive Protein (hs-CRP) | 6 weeks and 3 months
  Serum concentration of inflammatory marker high sensitive C-reactive Protein
Total fat tissue mass | 6 weeks and 3 months
  Total body fat mass measured with bioimpedance analysis
Lean tissue mass | 6 weeks and 3 months
  Lean tissue mass measured by bioimpedance analysis
Blood pressure | 6 weeks and 3 months
  Office measured blood pressure
Proteinuria | 6 weeks and 3 months
  Spot urinary protein to creatinine-ratio of the second morning urine
Serum potassium | 6 weeks and 3 months
  Serum potassium concentration (safety outcome)
Serum phosphate | 6 weeks and 3 months
  Serum phosphate concentration
Serum bicarbonate | 6 weeks and 3 months
  Serum concentration of bicarbonate (safety outcome)
Serum uric acid | 6 weeks and 3 months
  Serum uric acid concentration (safety outcome)
Micronutrient status of Selenium (safety outcome) | 6 weeks and 3 months
  Plasma Selenium concentration
n-3 Polyunsaturated Fatty Acid (PUFA) status | 6 weeks and 3 months
  n-3 PUFA content of erythrocyte lipid fraction
Urinary C-X-C motif chemokine 10 (CXCL10) | 6 weeks and 3 months
  Urinary levels of C-X-C motif chemokine 10 (CXCL10) as an indicator of tubulointerstital and microvascular inflammation
Gut produced uremic toxin p-cresyl sulphate | 6 weeks and 3 months
  Serum level of total and free p-cresyl sulphate
Urinary iodine concentration | 6 weeks and 3 months
  Urinary level of iodine concentration in ug/L
Plasma Zinc concentration (safety outcome) | 6 weeks and 3 months
  Plasma zinc concentration
Serum calcium concentration (safety outcome) | 6 weeks and 3 months
  Serum concentration of total calcium in mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Jernej Pajek, MD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baigent C, Landray MJ, Reith C, Emberson J, Wheeler DC, Tomson C, Wanner C, Krane V, Cass A, Craig J, Neal B, Jiang L, Hooi LS, Levin A, Agodoa L, Gaziano M, Kasiske B, Walker R, Massy ZA, Feldt-Rasmussen B, Krairittichai U, Ophascharoensuk V, Fellstrom B, Holdaas H, Tesar V, Wiecek A, Grobbee D, de Zeeuw D, Gronhagen-Riska C, Dasgupta T, Lewis D, Herrington W, Mafham M, Majoni W, Wallendszus K, Grimm R, Pedersen T, Tobert J, Armitage J, Baxter A, Bray C, Chen Y, Chen Z, Hill M, Knott C, Parish S, Simpson D, Sleight P, Young A, Collins R; SHARP Investigators. The effects of lowering LDL cholesterol with simvastatin plus ezetimibe in patients with chronic kidney disease (Study of Heart and Renal Protection): a randomised placebo-controlled trial. Lancet. 2011 Jun 25;377(9784):2181-92. doi: 10.1016/S0140-6736(11)60739-3. Epub 2011 Jun 12. PMID 21663949
- [Background] Barnard ND, Scialli AR, Turner-McGrievy G, Lanou AJ, Glass J. The effects of a low-fat, plant-based dietary intervention on body weight, metabolism, and insulin sensitivity. Am J Med. 2005 Sep;118(9):991-7. doi: 10.1016/j.amjmed.2005.03.039. PMID 16164885
- [Background] Van Breukelen GJ. ANCOVA versus change from baseline: more power in randomized studies, more bias in nonrandomized studies [corrected]. J Clin Epidemiol. 2006 Sep;59(9):920-5. doi: 10.1016/j.jclinepi.2006.02.007. Epub 2006 Jun 23. PMID 16895814
- [Background] Cartolano FC, Dias GD, de Freitas MCP, Figueiredo Neto AM, Damasceno NRT. Insulin Resistance Predicts Atherogenic Lipoprotein Profile in Nondiabetic Subjects. J Diabetes Res. 2017;2017:1018796. doi: 10.1155/2017/1018796. Epub 2017 Aug 22. PMID 28913361
- [Background] Claesson K, Mayer AD, Squifflet JP, Grabensee B, Eigler FW, Behrend M, Vanrenterghem Y, van Hooff J, Morales JM, Johnson RW, Buchholz B, Land W, Forsythe JL, Neumayer HH, Ericzon BG, Muhlbacher F. Lipoprotein patterns in renal transplant patients: a comparison between FK 506 and cyclosporine A patients. Transplant Proc. 1998 Jun;30(4):1292-4. doi: 10.1016/s0041-1345(98)00246-2. No abstract available. PMID 9636524
- [Background] Ferdowsian HR, Barnard ND. Effects of plant-based diets on plasma lipids. Am J Cardiol. 2009 Oct 1;104(7):947-56. doi: 10.1016/j.amjcard.2009.05.032. PMID 19766762
- [Background] Gardner CD, Coulston A, Chatterjee L, Rigby A, Spiller G, Farquhar JW. The effect of a plant-based diet on plasma lipids in hypercholesterolemic adults: a randomized trial. Ann Intern Med. 2005 May 3;142(9):725-33. doi: 10.7326/0003-4819-142-9-200505030-00007. PMID 15867404
- [Background] Heemann U, Abramowicz D, Spasovski G, Vanholder R; European Renal Best Practice Work Group on Kidney Transplantation. Endorsement of the Kidney Disease Improving Global Outcomes (KDIGO) guidelines on kidney transplantation: a European Renal Best Practice (ERBP) position statement. Nephrol Dial Transplant. 2011 Jul;26(7):2099-106. doi: 10.1093/ndt/gfr169. Epub 2011 May 9. PMID 21555392
- [Background] Holdaas H, Fellstrom B, Cole E, Nyberg G, Olsson AG, Pedersen TR, Madsen S, Gronhagen-Riska C, Neumayer HH, Maes B, Ambuhl P, Hartmann A, Staffler B, Jardine AG; Assessment of LEscol in Renal Transplantation (ALERT) Study Investigators. Long-term cardiac outcomes in renal transplant recipients receiving fluvastatin: the ALERT extension study. Am J Transplant. 2005 Dec;5(12):2929-36. doi: 10.1111/j.1600-6143.2005.01105.x. PMID 16303007
- [Background] Israni AK, Snyder JJ, Skeans MA, Peng Y, Maclean JR, Weinhandl ED, Kasiske BL; PORT Investigators. Predicting coronary heart disease after kidney transplantation: Patient Outcomes in Renal Transplantation (PORT) Study. Am J Transplant. 2010 Feb;10(2):338-53. doi: 10.1111/j.1600-6143.2009.02949.x. PMID 20415903
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Transplant Work Group. KDIGO clinical practice guideline for the care of kidney transplant recipients. Am J Transplant. 2009 Nov;9 Suppl 3:S1-155. doi: 10.1111/j.1600-6143.2009.02834.x. PMID 19845597
- [Background] Wanner C, Tonelli M; Kidney Disease: Improving Global Outcomes Lipid Guideline Development Work Group Members. KDIGO Clinical Practice Guideline for Lipid Management in CKD: summary of recommendation statements and clinical approach to the patient. Kidney Int. 2014 Jun;85(6):1303-9. doi: 10.1038/ki.2014.31. Epub 2014 Feb 19. PMID 24552851
- [Background] Lopes TS, Luiz RR, Hoffman DJ, Ferriolli E, Pfrimer K, Moura AS, Sichieri R, Pereira RA. Misreport of energy intake assessed with food records and 24-h recalls compared with total energy expenditure estimated with DLW. Eur J Clin Nutr. 2016 Nov;70(11):1259-1264. doi: 10.1038/ejcn.2016.85. Epub 2016 Jun 8. PMID 27273069
- [Background] Ojo AO, Hanson JA, Wolfe RA, Leichtman AB, Agodoa LY, Port FK. Long-term survival in renal transplant recipients with graft function. Kidney Int. 2000 Jan;57(1):307-13. doi: 10.1046/j.1523-1755.2000.00816.x. PMID 10620213
- [Background] Palmer SC, Navaneethan SD, Craig JC, Perkovic V, Johnson DW, Nigwekar SU, Hegbrant J, Strippoli GF. HMG CoA reductase inhibitors (statins) for kidney transplant recipients. Cochrane Database Syst Rev. 2014 Jan 28;2014(1):CD005019. doi: 10.1002/14651858.CD005019.pub4. PMID 24470059
- [Background] Prospective Studies Collaboration; Lewington S, Whitlock G, Clarke R, Sherliker P, Emberson J, Halsey J, Qizilbash N, Peto R, Collins R. Blood cholesterol and vascular mortality by age, sex, and blood pressure: a meta-analysis of individual data from 61 prospective studies with 55,000 vascular deaths. Lancet. 2007 Dec 1;370(9602):1829-39. doi: 10.1016/S0140-6736(07)61778-4. PMID 18061058
- [Background] Sniderman AD, Williams K, Contois JH, Monroe HM, McQueen MJ, de Graaf J, Furberg CD. A meta-analysis of low-density lipoprotein cholesterol, non-high-density lipoprotein cholesterol, and apolipoprotein B as markers of cardiovascular risk. Circ Cardiovasc Qual Outcomes. 2011 May;4(3):337-45. doi: 10.1161/CIRCOUTCOMES.110.959247. Epub 2011 Apr 12. PMID 21487090
- [Background] Authors/Task Force Members:; Catapano AL, Graham I, De Backer G, Wiklund O, Chapman MJ, Drexel H, Hoes AW, Jennings CS, Landmesser U, Pedersen TR, Reiner Z, Riccardi G, Taskinen MR, Tokgozoglu L, Verschuren WM, Vlachopoulos C, Wood DA, Zamorano JL. 2016 ESC/EAS Guidelines for the Management of Dyslipidaemias: The Task Force for the Management of Dyslipidaemias of the European Society of Cardiology (ESC) and European Atherosclerosis Society (EAS) Developed with the special contribution of the European Assocciation for Cardiovascular Prevention & Rehabilitation (EACPR). Atherosclerosis. 2016 Oct;253:281-344. doi: 10.1016/j.atherosclerosis.2016.08.018. Epub 2016 Sep 1. No abstract available. PMID 27594540